CLINICAL TRIAL: NCT05748795
Title: Microbial Colonization in Lung Cancer Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Tasneem Hassan Younes, Resident in chest department of assiut university hospital, Assiut University
Other Study IDs: Microbial colonization
Record Dates: First submitted 2023-01-23; First posted 2023-03-01 (Actual); Last update posted 2023-03-06 (Actual); Status verified 2023-02

CONDITIONS: Microbial Colonization
MeSH Terms: conditions — Communicable Diseases

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Biospecimen Retention: Samples Without DNA — * Bronchial wash and BAL will be processed within 2 h for bacterial, mycobacterial and mycological analysis using routine procedures. Specimens will be mixed and cultured on blood agar, chocolate agar, Sabarauds' Dextrose agar, MacConkey agar and Lowenstein Jensen medium.
  * Blood sample will be collected aseptically inoculated into the blood culture bottles, A blood culture system (BACT/ALERT 3D, BioMérieux Inc., Durham,USA) will be used for incubating blood culture samples and will be evaluated for 7 days. Positive blood culture bottles will be subjected to Gram's staining, cultured on blood agar, chocolate agar, Sabarauds' Dextrose agar and MacConkey agar.
  Bronchoscopic and blood culture samples that are positive for bacterial growth will undergo antimicrobial drug sensitivity testing .
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: bronchoscopy brochoalveolar lavage — * 2%lidocaine gel will be used to anaesthesize nasal mucosa.6ml lidocaine 2%diluted in 5cc normal saline lidocaine spray solution will be used for anaesthesizing the vocal cords and mucosa of the bronchial tree(13).
  * Intravenous midazolam (0.01-0.1mg\kg) will be given to achieve conscious sedation in selected cases(13).
  * Flexible Bronchoscopy will be done under continuous monitoring for O2 saturation, heart rate, blood pressure and respiratory rate.
  * The bronchoscope will be introduced into the nasal cavity and advanced to the level of the vocal cords. Lidocaine will be instilled through the bronchoscope to the vocal cords and tracheobronchial tree.
  * Using sterile bronchoscope in the lobar bronchus of tumor location,100 mL of sterile normal saline in fractionated doses will be injected and then BAL will be removed by suction to be collected in sterile side-way bottles.

SUMMARY:
Primary Aim:

-To determine the prevalence and pattern of bronchial colonization in patients presenting with lung cancer at the time of diagnosis

Secondary Aim:

-To assess the potential demographic, clinical, radiological and histological predictors of colonization in patients with lung cancer

DETAILED DESCRIPTION:
Lung cancer is the world's most common neoplasm and its incidence is rising. Lung cancer has the highest mortality rates of all cancers. Pulmonary infections, especially pneumonia, frequently complicate the course of lung cancer and are often the ultimate cause of death.

It has been suggested that bronchial colonization plays a key role in the establishment of pulmonary infections in patients with lung cancer, and thus clearly influences the therapeutic management and probably the prognosis of cancer.

In such patients, colonization may arise following local bronchial impairment, e.g. stenosis or impaired mucociliary clearance, or be caused by more general abnormalities, including immunosuppression, malnutrition, smoking, chronic obstructive pulmonary disease (COPD) and chemotherapy. Studies indicate that bronchial colonization can be demonstrated in 48.1% of patients with lung cancer and may be caused by potential pathogenic microorganisms (PPMs), mainly Haemophilus influenzae, Streptococcus pneumoniae and Staphylococcus aureus. Other potential microbial agents, such as mycobacteria and fungi, have not been investigated systematically However, there is a wide variation in the microbial profile reported from the previous studies; some of which reporting predominance of Gram-positive organisms- streptococcus pneumoniae in particular, while more recent studies reported predominance of Gram-negative organisms, which may indicate a shift in the spectrum of organism colonizing bronchial tree of lung cancer patients in parallel to the increased trends of antibiotic exposures, something this study will re-examine. Moreover, given the paucity of literature highlighting the potential predictors of colonization in such patients, overlooking data on radiological findings in lung cancer patients and underreporting the impact of comorbidities, this study aims to further explore a wider array of potential demographic, clinical, radiological and histological determinants.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Radiological findings on HRCT chest suggestive of lung cancer (lung mass, pulmonary nodules with , obstructive pneumonia, unexplained lung collapse, mediastinal lymphadenopathy)

Exclusion Criteria:

* Patients who demonstrate clinical, laboratory or radiological evidence of active pulmonary infection that requires antibiotic therapy
* Patients in whom histological evidence of lung cancer can't be proven after histopathology
* Patients deemed unfit for bronchoscopy

  * Uncorrected hypoxia under oxygen spo2 <90%
  * Uncontrolled cardiac arrhythmias despite medical treatment and arrhythmias associated with haemodynamic compromise .
  * patient who has risk factors for abnormal coagulation
  * Undrained Pneumothorax
  * Asthma and Chronic obstructive pulmonary disease who had suffered exacerbation during the preceding 3 weeks
  * Myocardial infarction in the previous 4 weeks

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study will be conducted on patients who are undergoing flexible bronchoscopy for diagnosis of Lung cancer. A written consent will be obtained from all participants prior to the procedure.
Sampling Method: Probability Sample
Enrollment: 103 (Estimated)
Dates: Start 2023-02-01 (Actual); Primary Completion 2024-02-01 (Estimated); Study Completion 2024-02-01 (Estimated)

PRIMARY OUTCOMES:
Prevalence of microbial colonization among the study population: | through the study completion , an average of 1 year
  Colonization will be defined as isolation of microorganisms from bronchoscopic wash samples at a threshold of 102 cfu.mL-1, whereas infection will be considered at .105 cfu.mL-1 . Regardless of the amount, isolation of mycobacteria and non-commensal fungi will be considered as colonization or an infection depending on the species isolated.
Predictors of microbial colonization among the study population: | through the study completion , an average of 1 year
  Demographic, clinical, radiological and histological data will be examined using univariate and multivariate regression analysis to identify their potential predictability of the colonization in patients with lung cancer.

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed M Abdelhadi, professor, Principal Investigator — Assiut University; Hebatallah G Rashed, professor, Principal Investigator — Assiut University
Locations (1):
- Tasneem Hassan Younes, Asyut, Egypt

REFERENCES:
- [Background] Chen W, Zheng R, Baade PD, Zhang S, Zeng H, Bray F, Jemal A, Yu XQ, He J. Cancer statistics in China, 2015. CA Cancer J Clin. 2016 Mar-Apr;66(2):115-32. doi: 10.3322/caac.21338. Epub 2016 Jan 25. PMID 26808342
- [Background] Gonzalez C, Johnson T, Rolston K, Merriman K, Warneke C, Evans S. Predicting pneumonia mortality using CURB-65, PSI, and patient characteristics in patients presenting to the emergency department of a comprehensive cancer center. Cancer Med. 2014 Aug;3(4):962-70. doi: 10.1002/cam4.240. Epub 2014 May 7. PMID 24802800
- [Background] D'Journo XB, Rolain JM, Doddoli C, Raoult D, Thomas PA. Airways colonizations in patients undergoing lung cancer surgery. Eur J Cardiothorac Surg. 2011 Aug;40(2):309-19. doi: 10.1016/j.ejcts.2010.11.036. Epub 2011 Jan 8. PMID 21216614
- [Background] Lanoix JP, Pluquet E, Lescure FX, Bentayeb H, Lecuyer E, Boutemy M, Dumont P, Jounieaux V, Schmit JL, Dayen C, Douadi Y. Bacterial infection profiles in lung cancer patients with febrile neutropenia. BMC Infect Dis. 2011 Jun 27;11:183. doi: 10.1186/1471-2334-11-183. PMID 21707992
- [Background] Laroumagne S, Salinas-Pineda A, Hermant C, Murris M, Gourraud PA, Do C, Segonds C, Didier A, Mazieres J. [Incidence and characteristics of bronchial colonisation in patient with lung cancer: a retrospective study of 388 cases]. Rev Mal Respir. 2011 Mar;28(3):328-35. doi: 10.1016/j.rmr.2010.05.020. Epub 2011 Feb 3. French. PMID 21482336
- [Background] Ioanas M, Angrill J, Baldo X, Arancibia F, Gonzalez J, Bauer T, Canalis E, Torres A. Bronchial bacterial colonization in patients with resectable lung carcinoma. Eur Respir J. 2002 Feb;19(2):326-32. doi: 10.1183/09031936.02.00236402. PMID 11866014
- [Background] 8. Zhou S, Zhao Q. Colonization of Streptococcus pneumoniae in Pneumonia Patients with Lung Cancer. Jundishapur Journal of Microbiology. 2018 Feb 28;11(2)
- [Background] 9. Stojanovic A. Bronchial Colonization in Patients with Non-Small Cell Lung Cancer. Acta Facultatis Medicae Naissensis. 2015 Apr 1;32(2):147.
- [Background] Laroumagne S, Lepage B, Hermant C, Plat G, Phelippeau M, Bigay-Game L, Lozano S, Guibert N, Segonds C, Mallard V, Augustin N, Didier A, Mazieres J. Bronchial colonisation in patients with lung cancer: a prospective study. Eur Respir J. 2013 Jul;42(1):220-9. doi: 10.1183/09031936.00062212. Epub 2012 Oct 25. PMID 23100491
- [Background] 11. Kirana WT, Desianti GA. Bacterial Colonizationin Lung Cancer Patients. InB68. CURIOUS PRESENTATIONS: CANCERS AND MIMICKERS 2022 May (pp. A3380-A3380). American Thoracic Society.
- [Background] Kang JY, Kang HS, Heo JW, Kim YH, Kim SJ, Lee SH, Kwon SS, Kim YJ. Clinical significance of microbial colonization identified by initial bronchoscopy in patients with lung cancer requiring chemotherapy. J Thorac Dis. 2021 Mar;13(3):1306-1314. doi: 10.21037/jtd-20-2722. PMID 33841924
- [Background] Du Rand IA, Blaikley J, Booton R, Chaudhuri N, Gupta V, Khalid S, Mandal S, Martin J, Mills J, Navani N, Rahman NM, Wrightson JM, Munavvar M; British Thoracic Society Bronchoscopy Guideline Group. British Thoracic Society guideline for diagnostic flexible bronchoscopy in adults: accredited by NICE. Thorax. 2013 Aug;68 Suppl 1:i1-i44. doi: 10.1136/thoraxjnl-2013-203618. No abstract available. PMID 23860341
- [Background] Feng SH, Yang ST. The new 8th TNM staging system of lung cancer and its potential imaging interpretation pitfalls and limitations with CT image demonstrations. Diagn Interv Radiol. 2019 Jul;25(4):270-279. doi: 10.5152/dir.2019.18458. PMID 31295144
- [Background] Ganti AKP, Loo BW, Bassetti M, Blakely C, Chiang A, D'Amico TA, D'Avella C, Dowlati A, Downey RJ, Edelman M, Florsheim C, Gold KA, Goldman JW, Grecula JC, Hann C, Iams W, Iyengar P, Kelly K, Khalil M, Koczywas M, Merritt RE, Mohindra N, Molina J, Moran C, Pokharel S, Puri S, Qin A, Rusthoven C, Sands J, Santana-Davila R, Shafique M, Waqar SN, Gregory KM, Hughes M. Small Cell Lung Cancer, Version 2.2022, NCCN Clinical Practice Guidelines in Oncology. J Natl Compr Canc Netw. 2021 Dec;19(12):1441-1464. doi: 10.6004/jnccn.2021.0058. PMID 34902832